CLINICAL TRIAL: NCT03975153
Title: An Open Label Pilot Trial of Guselkumab in the Treatment of Adults With Pityriasis Rubra Pilaris (PRP)
Brief Title: Guselkumab in the Treatment of Pityriasis Rubra Pilaris (PRP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Teri Greiling, Assistant Professor of Dermatology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00019343
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pityriasis Rubra Pilaris
Keywords: Interleukin-23, IL-23, guselkumab, Tremfya
MeSH Terms: conditions — Pityriasis Rubra Pilaris | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- guselkumab treatment (Experimental): Treatment with guselkumab for 20 weeks
  Interventions: Biological: guselkumab

INTERVENTIONS:
Biological: guselkumab — Treatment at the FDA-approved psoriasis dosing for 20 weeks
  Other Names: Tremfya

SUMMARY:
15 patients with PRP will be treated with guselkumab for 20 weeks to determine safety and efficacy. Participants are required to travel to Portland, OR only for the first visit, week-4 visit, and week-24 visit. 3 visits in between these times and one follow up visit may be performed by secure videoconferencing.

DETAILED DESCRIPTION:
Pityriasis rubra pilaris (PRP) is a rare and poorly understood severe inflammatory skin disease characterized by widespread (often full-body) redness and flaking of the skin, painful thickening and cracking of the palms and soles, hair loss, crumbling nails, and severe skin itching and burning.

There is no FDA-approved therapy for this rare disease and the commonly used medications do not work for many patients. There is some evidence that interleukin (IL)-23 may be too high in the skin of PRP patients. Ixekizumab is an injectable medication that blocks IL-23 by binding the p19 subunit and is FDA-approved for psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PRP by clinical assessment
* Male age 18-99, willing to use a reliable form of birth control if sexually active with a woman who is able to become pregnant.
* Female age 18-99; either of non-childbearing potential or of childbearing potential who test negative for pregnancy and agree to use a reliable method of birth control or remain abstinent during the study and for at least 12 weeks following the last dose of guselkumab.
* Involved body surface area (BSA) ≥ 10% at baseline (moderate-to-severe disease).
* Are a candidate for phototherapy and/or systemic therapy.

Exclusion Criteria:

* Willingness to travel to Oregon Health and Science University (OHSU) for all study visits, or willing/able to participate in remote videoconferencing visits with access to a computer with internet and webcam capabilities.
* Known malignancy or lymphoproliferative disease (except treated basal cell skin cancer, treated squamous cell skin cancer, or treated cervical carcinoma in situ) for at least 5 years.
* Active, untreated, acute or chronic infection, or immunocompromised to an extent that such that participation in the study would pose an unacceptable risk to the subject.
* Positive for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
* Have latent or active untreated tuberculosis (TB), a positive QuantiFERON-TB Gold test result, signs or symptoms of active TB on medical history or physical examination, or close contact with a person with active TB who have not undergone evaluation or treatment for TB. Those who are currently • Previous treatment with any agent that targets the interleukin 23 p19 subunit specifically.
* Systemic treatment with prednisone in the last 2 weeks, or other systemic therapies or phototherapy for PRP within the past 4 weeks or 5 half-lives prior to baseline, whichever is longer. For biologic therapies, the specific washout periods used will be: etanercept <28 days; infliximab, adalimumab, i
* Have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the subject if participating in this study.
* Have or intend to have a live vaccine within 3 months prior to baseline or 12 months prior to baseline in the case of the Bacillus Calmette-Guerin (BCG) vaccine, or any live vaccine during the course of study or within 3 months after the last administration of study drug.
* Had any major surgery within 8 weeks prior to baseline or will require major surgery during the study, that in the opinion of the investigator would pose an unacceptable risk to the subject.
* Presence of significant uncontrolled cerebrovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or neuropsychiatric disorders, or abnormal laboratory screening values that, in the opinion of the investigator, pose an unacceptable risk to the subject if participating • Have clinical laboratory test results at screening that are outside the normal reference range of the population and are considered clinically significant, or have any of the following specific abnormalities: Neutrophil count <1500 cells/μL, white blood cell count <3500 cells/μL, platelet count <100,000
* Women who are lactating or breastfeeding.
* Have any other condition that precludes the subject from following and completing the protocol, in the opinion of the investigator.
* Are investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child, or sibling).
* Are currently enrolled in, or discontinued from a clinical trial involving an investigational product or non-approved use of a drug or device within the last 4 weeks or a period of at least 5 half-lives of the last administration of the drug, whichever is longer, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teri Greiling, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Velasco RC, Shao C, Cutler B, Strunck J, Kent G, Cassidy PB, Choate K, Greiling TM. Guselkumab for Pityriasis Rubra Pilaris and Dysregulation of IL-23/IL-17 and NFkB Signaling: A Nonrandomized Trial. JAMA Dermatol. 2024 Jun 1;160(6):641-645. doi: 10.1001/jamadermatol.2024.0257. PMID 38598229

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guselkumab Treatment
Started | 14
Completed | 12
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Per-protocol population
Arm/Group | Guselkumab Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Psoriasis Area and Severity Index [Mean (Standard Deviation); unit: units on a scale] — Measures the appearance of the skin based on erythema, scale, and elevation, multiplied by body surface area. 0 indicates completely clear skin. 72 is the maximum value, indicating the worst severity. A score of 11 or higher is considered severe disease.
  units on a scale | 30.6 (11.4)
Dermatology Life Quality Index [Mean (Standard Deviation); unit: units on a scale] — The DLQI is calculated by adding the score for 10 questions, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
  units on a scale | 20.1 (6.8)
Itch numeric rating scale [Mean (Standard Deviation); unit: units on a scale] — Participants are asked to rate their average itch in the last 2 weeks on a 0 to 10-point scale, with 0 being no itch and 10 being the worst itch imaginable.
  units on a scale | 6.9 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Psoriasis Area and Severity Index (PASI) at Week-24 After Treatment With Guselkumab.
Description: PASI measures the appearance of the skin based on erythema, scale, and elevation, multiplied by body surface area. 0 indicates completely clear skin. 72 is the maximum value, indicating the worst severity. A score of 11 or higher is considered severe disease.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: percent change from baseline PASI
Arm/Group | Guselkumab Treatment
Number analyzed (Participants) | 12
percent change from baseline PASI | 61.8 [21.3 to 100]

2. Secondary Outcome: Proportion of Subjects Achieving a 4-point Improvement in Quality of Life Measured by the Dermatology Life Quality Index (DLQI) at Week-24.
Description: Quality of life will be measured by the Dermatology Life Quality Index (DLQI). There are 10 questions covering symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question refers to the impact of PRP on the patient's life over the previous week. The highest score is 30 and would indicate a maximum (negative) impact on quality of life. A score of zero would indicate no impact on quality of life. For inflammatory skin conditions, a 4-point improvement in DLQI score is considered clinically important.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab Treatment
Number analyzed (Participants) | 12
Participants | 11

3. Secondary Outcome: Proportion of Subjects With >50% Improvement With Psoriasis Area and Severity Index (PASI) at Week-24 Who Did Not Worsen at Week-36
Description: PASI measures the appearance of the skin based on erythema, scale, and elevation, multiplied by body surface area. 0 indicates completely clear skin. 72 is the maximum value, indicating the worst severity. A score of 11 or higher is considered severe disease. Trial participants who had a decrease in PASI by >50% from week-0 to week-24 were included in this analysis. Participants did not receive any additional doses of guselkumab after week-20, and PASI score at week-36 was calculated to assess for sustained remission.
Time Frame: 36 weeks
Population: Only participants who achieved >50% in PASI at week-24 are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab Treatment
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Guselkumab Treatment
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guselkumab Treatment (N=12)
Cholecystitis leading to myocardial infarction and death (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guselkumab Treatment (N=12)
Temporary PRP worsening (Skin and subcutaneous tissue disorders) | 1 (1)
Ectropion (Eye disorders) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Ground level fall (Social circumstances) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pustules (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
False-positive hyperkalmia (Blood and lymphatic system disorders) | 1 (1)
COVID19 infection (Infections and infestations) | 1 (1)
Type 2 diabetes (Endocrine disorders) | 1 (1)
Bell's palsy (Nervous system disorders) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 1 (1)
Leukocytosis (Immune system disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Fall due to plantar fissures (General disorders) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1)
Ruptured blister (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the study: open label design, small sample size, lack of validated outcomes measures for PRP, racial and ethnic homogeneity of the participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT03975153/Prot_SAP_000.pdf